CLINICAL TRIAL: NCT06066814
Title: To Study the Role of Plasma Von Willebrand Factor Antigen (vWF) to A Disintegrin-like and Metalloproteinase With Thrombospondin Type-1 Motifs 13 (ADAMTS-13) Activity Ratio as a Predictor of Development of Extrahepatic Organ Failure in Acute on Chronic Liver Failure (ACLF) Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-ACLF-14
Record Dates: First submitted 2023-09-28; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Acute on Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute on chronic liver failure (ACLF) is a syndrome characterized by acute decompensation of chronic liver disease associated with organ failures and high short- term mortality. Development of systemic inflammation and subsequent organ failures determines is associate with poor outcome and short-term mortality. Previous studies have shown that endothelial injury leading to increase in levels of and exhaustion of its cleaving protein a disintegrin and metalloproteinase with a thrombospondin type 1 motif, member 13 (ADAMTS 13) which promotes the platelet microthrombi formation and subsequent organ ischemia. We propose that the vWF : ADAMTS 13 ratio can be predict the organ failure development and subsequent mortality in ACLF patients, which is considered to be a inflammatory state.

DETAILED DESCRIPTION:
Null Hypothesis:

Systemic inflammation in acute-on-chronic liver failure (ACLF) leads to endothelial injury leading to increased vWF levels and exhaustion of its cleaving protein ADAMTS 13 which promotes the platelet microthrombi formation, leading to subsequent organ failures which are the strong predictors of short term mortality.

AIM: - To evaluate the role of plasma Von Willebrand factor antigen to ADAMTS-13 activity ratio in predicting organ failure in acute on chronic liver failure (ACLF) patients Objective -

Primary objective:

To study efficacy of Von Willebrand factor antigen to ADAMTS-13 activity ratio in predicting development of organ failures at day 7

Secondary objectives:

1. To study efficacy of vWF Ag : ADAMTS-13 ratio in predicting 28 days transplant free survival.
2. To study efficacy of day 1 and day 4 vWF and ADAMTS 13 level with in predicting development of organ failures at day.
3. To efficacy of day 1 and day 4 vWF and ADAMTS 13 level with in predicting 28 days transplant free survival.
4. To compare vWF, ADAMTS 13 level and vWF Ag : ADAMTS-13 ratio across different grades of AARC ACLF.
5. To compare vWF, ADAMTS 13 level and vWF Ag : ADAMTS-13 ratio with AARC, MELD, SOFA, CLIF-ACLF scores.
6. To compare the impact of different therapies on vWF, ADAMTS 13 level and vWF Ag : ADAMTS-13 ratio (PLEX, Etiology specific : steroids, antivirals).

Study population: All the patients with age >18 years who are diagnosed having ACLF fulfilling APASL ACLF criteria Study design: Prospective cohort study Study period: September 2023 - December 2023 Intervention: This is a prospective cohort study and will be conducted at ILBS New Delhi

The following data will be recorded for each patient:

H/o of jaundice, distension abdomen, swelling feet, altered sensorium, vomiting of blood or passing melena Acute and chronic etiology of ACLF Clinical examination: Ascites with grade, glass glow coma scale, west heaven hepatic encephalopathy grade, heart rate, blood pressure, urine output Height, weight and BMI Day 0 - Routine investigations: Hemogram, TLC, DLC, KFT, LFT, Prothrombin time/INR D-Dimer, Fibrinogen, ROTEM, arterial lactate Von Willebrand factor antigen, ADAMTS 13 activity Organ failure assessment with SOFA score Disease Severity assessment with AARC/MELD/CLIF-ACLF DAY 4 - Routine investigations: Hemogram, TLC, DLC, KFT, LFT, Prothrombin time/INR D-Dimer, Fibrinogen, ROTEM, arterial lactate Von Willebrand factor antigen, ADAMTS 13 activity Organ failure assessment with SOFA score Disease Severity assessment with AARC/MELD/CLIF-ACLF DAY 7: - Routine investigations: Hemogram, TLC, DLC, KFT, LFT, Prothrombin time/INR D-Dimer, Fibrinogen, ROTEM, arterial lactate Von Willebrand factor antigen, ADAMTS 13 activity Organ failure assessment with SOFA score Disease Severity assessment with AARC/MELD/CLIF-ACLF Day 28- Final outcome assessment death or alive Total five organs parameters will be assessed: Kidney, Brain, Coagulation, Circulatory, Respiratory

Liver failure will be assessed by AARC score:

Extrahepatic organ failure/dysfunction will be assessed by CLF SOFA score

Organ failure will be defined as:

Renal failure: Creatinine >2.0 mg/dL or RRT Cerebral failure: Grade 3-4 Circulatory failure: Vasopressor requirement Respiratory failure: PaO2/FiO2 <200 or SpO2/FiO2 <214 Monitoring and assessment: All the parameters of the objective and also noted any adverse effects.

STATISTICAL ANALYSIS:

The data will be entered in Microsoft excel and will be analyzed using SPSS version 22. The categorical data will be analysed using Chi square/Fissure test. Exact test and continuous data will be compiled using t-test. Besides this the univariate and multivariate survival analysis will be carried out using Cox regression method. Kaplan-Meier technique will be applied for further analysis. P-value<0.05 will be considered as significant.

Adverse effects: NA

ELIGIBILITY:
Inclusion Criteria:

- All the patients with age >18 years who are diagnosed having ACLF fulfilling APASL ACLF criteria and do not have any extrahepatic organ failure at enrollment.

Exclusion Criteria:

1. Patients on antiplatelet or anticoagulant therapy for at any point of time in last 7 days
2. Pregnant female
3. Patient receiving N-acetyl cysteine (NAC) (interferes with the vWF assay)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients with age >18 years who are diagnosed having ACLF fulfilling APASL ACLF criteria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-07 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients developing of any organ failures by day 7 with increased vWF: ADAMTS 13 ratio | Day 7

SECONDARY OUTCOMES:
Proportion of patients alive by day 28 without transplant with increased vWF: ADAMTS 13 ratio. | Day 28
Proportion of patients developing of any organ failures by day 7 with increased day 1 and day 4 vWF and ADAMTS 13 level. | Day 7
Proportion of patients alive by day 28 without transplant with increased day 1 and day 4 vWF and ADAMTS 13 level. | Day 28
Proportion of patients with increased vWF, ADAMTS 13 level and vWF Ag : ADAMTS-13 ratio across different grades of AARC ACLF | Day 28
Proportion of patients having change in vWF, ADAMTS 13 level and vWF Ag : ADAMTS-13 ratio compared to change in AARC, MELD, CLIF-ACLF scores | Day 28
Proportion of patients having change in vWF, ADAMTS 13 level and vWF Ag : ADAMTS-13 ratio at day 7 different therapies (Nutrition, Plasma exchange, Prednisolone, Nucleos(t)ide analogue in hepatitis B) on vWF, ADAMTS 13 level and vWF Ag : ADAMTS-13 ratio. | Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences., New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided